CLINICAL TRIAL: NCT04071821
Title: A Randomized, Open-Label, Single-Dose, Five-Period Crossover, Relative Bioavailability Study to Evaluate Cetirizine HCl Gummy 10 mg and Cetirizine HCl Oral Tablets 10 mg Administered in Healthy Adult Male and Female Subjects
Brief Title: Relative Bioavailability Study to Evaluate Cetirizine HCl Gummy 10 mg and Cetirizine HCl Oral Tablets 10 mg
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Gummy Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P001-2019
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Cetirizine

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, Single-Dose, Five-Period Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- A: Test under Fasted Condition (Experimental): Single oral dose of cetirizine HCl Gummy 10 mg, chewed, administered with approximately 240 mL of room temperature water, under fasted conditions
  Interventions: Drug: cetirizine HCl Gummy
- B: Reference under Fasted Condition (Active Comparator): Reference: Single oral dose of cetirizine HCl oral tablets 10 mg, administered with approximately 240 mL of room temperature water, under fasted conditions
  Interventions: Drug: Zyrtec tablet 10mg
- C: Test under Fed Condition (Experimental): Test: Single oral dose of cetirizine HCl Gummy 10 mg, chewed, administered with approximately 240 mL of room temperature water, under fed conditions
  Interventions: Drug: cetirizine HCl Gummy
- D: Test under Fasted Condition with No Water (Experimental): Single oral dose of cetirizine HCl Gummy 10 mg, chewed, administered with no water, under fasted conditions
  Interventions: Drug: cetirizine HCl Gummy
- E: Test Swallowed Whole with Water, under Fasted Condition (Experimental): Single oral dose of cetirizine HCl Gummy 10 mg, swallowed whole, administered with approximately 240 mL of room temperature water, under fasted conditions
  Interventions: Drug: cetirizine HCl Gummy

INTERVENTIONS:
Drug: cetirizine HCl Gummy — cetirizine HCl 10mg in a gummy formulation
  Other Names: Ceteric Allergy Gummy
  Arms: A: Test under Fasted Condition; C: Test under Fed Condition; D: Test under Fasted Condition with No Water; E: Test Swallowed Whole with Water, under Fasted Condition
Drug: Zyrtec tablet 10mg — cetirizine HCl 10mg tablet
  Arms: B: Reference under Fasted Condition

SUMMARY:
A Randomized, Open-Label, Single-Dose, Five-Period Crossover, Relative Bioavailability Study to Evaluate Cetirizine HCl Gummy 10 mg and Cetirizine HCl Oral Tablets 10 mg Administered in Healthy Adult Male and Female Subjects

DETAILED DESCRIPTION:
Primary:

• To determine the relative bioavailability of a single oral dose of cetirizine HCl Gummy 10 mg and cetirizine HCl oral tablets 10 mg administered under fasted conditions in healthy adult male and female subjects.

Secondary:

* To determine the relative bioavailability of a single oral dose of cetirizine HCl Gummy 10 mg administered under fasted and fed conditions in healthy adult male and female subjects;
* To determine the relative bioavailability of a single oral dose of cetirizine HCl Gummy 10 mg administered under fasted conditions with and without water in healthy adult male and female subjects;
* To determine the relative bioavailability of a single oral dose of cetirizine HCl Gummy 10 mg administered under fasted conditions and chewed or swallowed whole in healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of giving informed consent and complying with study procedures;
2. Male or female, 18 to 55 years of age, inclusive, at date of consent;
3. Body mass index (BMI) ≥ 18.0 to ≤ 32.0 kg/m2 and total body weight > 50 kg (110 lbs.) at Screening;
4. All female subjects must have a negative pregnancy test at Screening and at each Check-in Visit; and one of the following:

   1. Using a medically acceptable form of birth control for at least 1 month prior to first dose [e.g., hormonal contraceptives (oral, patch, injectable or vaginal ring), intrauterine device, or a double barrier method (e.g., diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge)]
   2. Documented as surgically sterile by hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/tubal occlusion) at least 6 months prior to the first dose;
   3. Postmenopausal (no menstruation for a minimum of 12 months and confirmed by FSH and estradiol at Screening);
5. Medically healthy based on medical history, vital sign measurements, clinical laboratory test results, and physical examination;
6. Non-smokers (including nicotine-containing products) for at least 6 continuous months prior to the first dose.
7. Be willing and able to consume all contents of the standardized high calorie, high fat breakfast within 30 minutes prior to dosing.

Exclusion Criteria:

1. Females who are pregnant, lactating, or planning to become pregnant during the study;
2. Life-time history and/or recent evidence of alcohol or drug/substance abuse disorder;
3. Subjects with history of hypersensitivity to cetirizine or hydroxyzine, or any component of the test and reference formulations;
4. Subjects who test positive at Screening for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody;
5. Subjects who test positive at Screening or at Check-in for alcohol and/or drugs of abuse;
6. Subjects who donated ≥ 500 mL of blood within 56 days prior to the first dose of study drug or ≥ 50 mL and ≤ 499 mL of blood within 30 days or plasma (e.g. plasmapheresis) within 14 days prior to the first dose of study drug;
7. Use of prescription or non-prescription drugs, dietary supplements, or herbal supplements at the time of Screening and within 14 days prior to the first dose of the study drug;
8. Subjects who have a history of difficulty in donating blood or difficulty with phlebotomy procedures, and poor venous access;
9. Subjects who have participated in another clinical trial within 30 days prior to the first study period;
10. Member or first-degree relative of study staff or the Sponsor directly involved in the study;
11. Any condition which in the opinion of Investigator would interfere with the subject's ability to provide informed consent, comply with study instructions, confound interpretation of study results, or endanger the subject if he or she took part in the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
maximum plasma cetirizine concentration (Cmax) | 2 months
  PK blood samples to measure plasma concentrations of cetirizine will be collected by direct venipuncture or by use of an indwelling cannula. Blood will be collected into tubes containing K2EDTA for determination of plasma cetirizine concentration at time 0 (within 60 minutes pre-dose), 10, 20 minute post-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36 hours post-dose. Plasma cetirizine concentrations will be listed at each time point by subject and summarized by treatment at each time point using descriptive statistics (n, mean, standard deviation (SD), Coefficient of variation (CV%), median, minimum and maximum values). Pharmacokinetic calculations will be performed based on actual time of blood sample collection, using non-compartmental methods with Phoenix WinNonlin Version 8.1 (Certara USA, Inc., Princeton, New Jersey, USA). Plots of mean concentrations of plasma cetirizine versus time will be generated and Cmax will be generated from the plot.
area under the plasma drug concentration versus time curve (AUC) | 2 months
  AUC will be determined using non-compartmental analysis methods (Phoenix WinNonlin software, version 8.1 or higher, Certara USA Inc., Princeton, NJ). AUC will be calculated to the last measurable observation (AUC0-t) and extrapolated to infinity (AUC0 ∞).

SECONDARY OUTCOMES:
time to Cmax (Tmax) | 2 months
  Tmax will be determined using non-compartmental analysis methods (Phoenix WinNonlin software, version 8.1 or higher, Certara USA Inc., Princeton, NJ).
elimination half-life (t½) | 2 months
  t½ will be determined using non-compartmental analysis methods (Phoenix WinNonlin software, version 8.1 or higher, Certara USA Inc., Princeton, NJ).
terminal elimination rate constant (Kel). | 2 months
  Kel will be determined using non-compartmental analysis methods (Phoenix WinNonlin software, version 8.1 or higher, Certara USA Inc., Princeton, NJ).

OTHER OUTCOMES:
incidence of treatment-emergent adverse events (TEAE) | 2 months
  Adverse events (AE) will be coded using a standardized Medical Dictionary for Regulatory Activities (MedDRA), Version 22,0 or higher. All treatment-emergent adverse events (TEAE) will be documented throughout the study from the time a subject receives the first dose of study drug until 7 days after the subject receives the last dose of study drug.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-07-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT04071821/Prot_000.pdf